CLINICAL TRIAL: NCT04516785
Title: Reducing Colonoscopies in Patients Without Significant Bowel Disease
Acronym: RECEDE
Status: Completed | Type: Observational
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Collaborators: University of Warwick (Other); University of Leeds (Other); University of Manchester (Other)
Responsible Party: Sponsor
Other Study IDs: RA481020
Record Dates: First submitted 2020-08-13; First posted 2020-08-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Colorectal Cancer; Colorectal Disorders; Colorectal Adenoma; Colorectal Polyp
Keywords: gastroenterology; colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention: FIT and urine VOC samples followed by colonoscopy
  Interventions: Diagnostic Test: FIT and VOC

INTERVENTIONS:
Diagnostic Test: FIT and VOC — Stool sample (FIT) analysed for blood in faeces and urine sample (VOC) analysed for the presence of volatile organic compounds

SUMMARY:
Investigating people with bowel symptoms uses a test that detects traces of blood in the stools, the FIT test. There are many possible reasons for positive tests. A few people have cancer. However, most participants with symptoms don't have any serious bowel disease but have benign problems such as piles or irritable bowel syndrome (IBS). It is very difficult to diagnose on symptoms alone, those participants who have serious bowel disease and those who do not.

After a positive test, people are invited for colonoscopy - a sort of articulated tube that is passed up the bowel. Most people invited for colonoscopy don't have cancer. Only about 5% of those with positive FIT tests have cancer. About 25% have other bowel diseases, but most have nothing serious wrong at all. So they have the inconvenience and discomfort of colonoscopy but don't get any benefit from it.

The investigators want to try adding another test, the volatile organic compound (VOC) test, to see if the investigators can separate those with positive FIT tests who do have something wrong, from those who don't. The VOC test uses a urine sample. Using both tests might also be better for detecting cancer. FIT alone misses about 20%.

So the investigators think that using both tests might not only be better for detecting cancer, but also might mean that a lot of people will avoid having to have colonoscopy.

This study will recruit 1,819 participants with bowel symptoms from NHS trusts in the UK. They will provide stool samples for FIT and urine for VOC analysis. They will have colonoscopy to get a definite diagnosis. Then the investigators will look at their FIT and VOC test results to see if in future, people with both tests negative.

DETAILED DESCRIPTION:
There is currently disparity between demand and available resources for colonoscopy. At present around 300,000 participants (and rising) are being referred annually to NHS trusts suspected of colorectal cancer (CRC). These participants are offered invasive colonic examinations (colonoscopy or CT colonography) but only 30% will have significant bowel disease. Significant bowel disease includes neoplasia (cancer and benign tumours) and significant treatable benign conditions such as inflammatory bowel disease and microscopic colitis. Of the remaining 70%, 40% have completely normal colonic investigations and 30% have functional bowel conditions such as irritable bowel syndrome or diverticular disease.

Set against this there is and will remain for the foreseeable future a capacity shortfall for colonoscopy. This limits the ability of the NHS to extend colorectal cancer detection within the Bowel Cancer Screening Programme (BCSP) or to target those participants that present for the first time through the Emergency Department (25% of all colorectal cancer diagnoses).

The increasing demand, limited capacity and lack of a triage tests have left NHS trusts with a conundrum of how best to stratify those with symptoms and at risk of SBD including CRC. The National Institute for Health and Care Excellence (NICE) has recommended a stool test (faecal immunochemical testing for haemoglobin, known as FIT) in the assessment of those suspected of CRC. NICE have recommended 10 μgHb/g faeces as the cut off for investigation of people with low risk symptoms who, account for only 10% of those referred with suspected CRC. When applied to high risk symptom groups, FIT will miss a significant number of participants with CRC (~10%) if used on its own at the threshold recommended by NICE (10 μgHb/g faeces). FIT will also miss a large number of significant potentially pre-cancerous polyps (~40%). Early detection and removal of such polyps will reduce risk of CRC.

The Bowel Cancer Screening Programme (BCSP) has set a FIT cut off of >120 μgHb/g faeces, compared to the NICE threshold of 10 μgHb/g faeces, but even at the lower threshold recommended by NICE some SBDs will be missed. Whilst a lower threshold might improve detection of SBD, it will increase the number of colonoscopies that find no abnormality. Consequently, the investigators have been investigating a urine test (in addition to FIT) to improve detection of participants with SBD with a view to reducing unnecessary colonoscopies. The urine test analyses volatile organic compounds (VOCs) that originate from the body and provides a chemical 'fingerprint' that is disease specific. Stool FIT and urine VOCs identify different biological characteristics of SBD - haemoglobin (as a marker of excess blood loss) versus metabolic response to inflammation. In a preliminary study of 562 participants, stool FIT on its own (at a threshold determined from the data) detected 80% of those with colorectal cancer. However, the addition of urine chemical testing improved this to 97%. The number of CRC cases missed by combined FIT and urine chemical testing is similar to that of colonoscopy, the current gold standard.

ELIGIBILITY:
Inclusion Criteria:

* - All participants referred either routinely with lower gastrointestinal symptoms or urgently (fulfilling the national criteria for referral - NICE NG12) for colonoscopy investigation that is determined by their overseeing clinician
* Minimum age of 18
* Able to provide informed consent
* Have the ability to return both stool and urine samples

Exclusion Criteria:

* Those who are pregnant

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants referred either routinely with lower gastrointestinal symptoms or urgently (fulfilling the national criteria for referral - NICE NG12) for colonoscopy investigation that is determined by their overseeing clinician
Sampling Method: Non-Probability Sample
Enrollment: 1181 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of stool FIT plus urine VOC compared to stool FIT alone to improve detection of SBD. | 24 months
  Sensitivity, specificity, negative predictive value (NPV) and positive predictive value (PPV) of stool FIT plus urine VOC in detection of SBD, using colonoscopy histology findings.

SECONDARY OUTCOMES:
Diagnostic accuracy of stool FIT plus urine VOC in detection of SBD | 24 months
  Receiver operating characteristic (ROC) curve of stool FIT plus urine VOC in detection of SBD to optimise the detection threshold.
Impact on number of colonoscopies undertaken | 24 months
  Calculation of potential number of colonoscopies avoided in those without SBD.
Cost effectiveness and colonoscopy disutility | 24 months
  Cost calculation, Quality of life (EQ-5D-5L) and quality adjusted life years (QALY) associated with utility of each diagnostic strategy (stool FIT and urine VOC) will be assessed to create a model that will employ a multi-part structure, consisting of a decision tree to evaluate short-term cost and consequences accruing at the diagnosis stage followed by a state-transition model to capture the long-term (lifetime) outcomes associated with the diagnosed condition.

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - University Hospital Coventry and Warwickshire NHS Trust, Coventry, West Midlands
  - University Hospital Derby & Burton, Derby
  - East Cheshire NHS Trust, Macclesfield
  - Milton Keynes University Hospital, Milton Keynes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bradley C, Hee SW, Andronis L, Persaud K, Hull MA, Todd J, Taylor-Phillips S, Smith S, Constable R, Waugh N, Arasaradnam RP; RECEDE Study Group. REducing Colonoscopies in patients without significant bowEl DiseasE: the RECEDE Study - protocol for a prospective diagnostic accuracy study. BMJ Open. 2022 Mar 30;12(3):e058559. doi: 10.1136/bmjopen-2021-058559. PMID 35354626